CLINICAL TRIAL: NCT03347500
Title: Development of a Microfluidic Organotypic Model to Evaluate Monocyte Transendothelial Migration to the Joint in Obese Osteoarthritic Patients
Brief Title: Microfluidic Organotypic Model for Monocyte Transendothelial Migration to the Joint in Obese Osteoarthritic Patients
Acronym: MOTEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: MOTEM
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese OA patients: Use of patient-derived biological samples
  Inclusion Criteria:
  * Subscription of informed consent
  * BMI ≥ 30
  * age between 60-80 years included
  * Kelgrenn-Lawrence equal or superior to grade III
  * presence of synovitis
  * patients undergoing knee replacement
  * suspension of NSAIDs from one week before the surgical procedure according to the standard clinical practice
  Exclusion criteria:
  - HCV, HIV, HBV, TPHA infection
  Interventions: Other: use of patient-derived biological samples
- Non-obese OA patients: Use of patient-derived biological samples
  Inclusion criteria:
  * Subscription of informed consent
  * BMI ≤ 28
  * age between 60-80 years included
  * Kelgrenn-Lawrence equal or superior to grade III
  * presence of synovitis
  * patients undergoing knee replacement
  * suspension of NSAIDs from one week before the surgical procedure according to the standard clinical practice
  Exclusion criteria:
  - HCV, HIV, HBV, TPHA infection
  Interventions: Other: use of patient-derived biological samples

INTERVENTIONS:
Other: use of patient-derived biological samples — We will use biological samples that are routinely collected as waste material from patients undergoing prosthetic surgery at IRCCS Istituto Ortopedico Galeazzi. Peripheral blood will be also collected from patients during the pre-surgery visit and during the post-surgery hospitalization coinciding with routine blood sample collection.

SUMMARY:
Osteoarthritis (OA) is the fastest growing cause of disability worldwide due to population ageing and increasing obesity incidence. Obese individuals have a higher risk of OA insurgence and severe progression due to several risk factors, including their systemic inflammation state and superior migratory ability of monocytes. In the present project we aim at the development of a novel 3D microfluidic organotypic model resembling the joint to investigate the migration ability of monocytes from obese and non-obese OA patients.

We hypothesize that monocytes from obese OA patients display superior migration ability and a specific pattern of chemokine surface receptors compared to monocytes from non-obese OA patients. We also hypothesize that these features lead to a superior infiltration of monocytes/macrophages to the synovial membrane in obese OA patients. Based on this, our main aim will be to highlight differences between Mo from obese and non-obese OA patients in terms of surface receptors and migration ability in a microfluidic organotypic model.

ELIGIBILITY:
Inclusion criteria

Obese OA patients

* Subscription of informed consent
* BMI ≥ 30
* age between 60-80 years included
* Kelgrenn-Lawrence equal or superior to grade III
* presence of synovitis
* patients undergoing knee replacement
* suspension of NSAIDs from one week before the surgical procedure according to the standard clinical practice

Non-obese OA patients

* Subscription of informed consent
* BMI ≤ 28
* age between 60-80 years included
* Kelgrenn-Lawrence equal or superior to grade III
* presence of synovitis
* patients undergoing knee replacement
* suspension of NSAIDs from one week before the surgical procedure according to the standard clinical practice

Exclusion criteria

Obese OA patients - HCV, HIV, HBV, TPHA infection

Non-obese OA patients

- HCV, HIV, HBV, TPHA infection

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OA patients undergoing prosthetic surgery at IRCCS Istituto Ortopedico Galeazzi
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Chemokine receptor expression | 24 hours
  To evaluate and compare the expression of chemokine surface receptors on monocytes from obese and non-obese OA patients.

SECONDARY OUTCOMES:
Monocyte transendothelial migration | 48 hours
  To monitor the transendothelial migration of monocytes from OA patients in response to chemokines present in the synovial fluid using a microfluidic organotypic model.